CLINICAL TRIAL: NCT06629935
Title: Assessment of How Different Instrument Modifications in Le Fort I Surgery Influence the Osteotomy of the Lateral Nasal Wall, With a Focus on the Level of Fractures and the Separation Pattern of the Pterygomaxillary Junction
Brief Title: Impact of Different Instrument Modifications on Lateral Nasal Wall Osteotomy and Pterygomaxillary Separation in Le Fort I Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-KAEK-03
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Le Fort; I; Blood Loss
Keywords: orthognthic surgery; le fort I; lateral nasal wall; pterygomaxillary junction
MeSH Terms: conditions — Hemorrhage | interventions — Orthognathic Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nievert osteotomy group (Experimental): lateral nasal wall osteotomy has been performed with single guided Nievert osteotome.
  Interventions: Procedure: orthognathic surgery
- Blade osteotomy group (Active Comparator): lateral nasal wall osteotomy has been performed with blade osteotome.
  Interventions: Procedure: orthognathic surgery

INTERVENTIONS:
Procedure: orthognathic surgery — Le Fort I surgery

SUMMARY:
The aim of this study is to investigate the effect of different instrument modifications on the customized osteotomy of the lateral nasal wall in Le Fort I surgery, focusing on the level of lateral nasal wall fractures and the separation pattern of the pterygomaxillary junction.

The primary hypothesis is blade osteotome is useful and facilitate the fracture line in ideal level both for lateral nasal wall and the pterygomaxillary junction.

DETAILED DESCRIPTION:
While there are numerous studies in the literature evaluating various parameters related to maxillary down-fracture in Le Fort I osteotomy, studies specifically focused on lateral nasal osteotomy are very rare. There is no study in the literature has addressed customized lateral nasal osteotomy using different instruments. In our study, the lateral nasal wall osteotomy will be performed 2 mm shorter than the measured descending palatine ater distance in the axial computer tomography plane. One group (n=23) will use the routinely employed Nievert osteotome (single guided osteotome), while the other group (n=23) will use a blade osteotome (no guided tip). This study aims to evaluate parameters such as the fracture pattern of the lateral nasal walls and the separation pattern of the pterygomaxillary junction by using different instrument modifications for lateral nasal wall osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring Le Fort I or bimaxillary surgery
* Patients who have not previously undergone Le Fort I or bimaxillary surgery (revision)
* Patients without cleft lip or palate
* Patients with no history of midface fractures or craniofacial trauma

Exclusion Criteria:

* Patients with cleft lip and/or palate requiring orthognathic surgery
* Patients with a history of trauma needing orthognathic surgery for malocclusion correction
* Patients who have previously undergone orthognathic surgery and require revision surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
lateral nasal wall fracture type | 6 months
  Class 1: Fracture at the osteotomy line Class 2: Fracture 2-4 mm above the osteotomy line Class 3: Fracture more than 4 mm above the osteotomy line

SECONDARY OUTCOMES:
pterygomaxillary junction fracture type | 6 months
  Class 1: Separation at the tuberosity of the maxilla Class 2: Separation at the pterygomaxillary junction Class 3: Separation of the pterygoids plates

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No